CLINICAL TRIAL: NCT06232356
Title: Respiratory Health Screening Using a Mobile Device
Brief Title: Screening for Lung Health by a Mobile Device
Acronym: SMILE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SEPAR- EPOC (Other)
Responsible Party: Sponsor
Other Study IDs: SAP_SMILE_2864995
Record Dates: First submitted 2024-01-18; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Lung Diseases; COPD
Keywords: Spirometry
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: The study population will consist of adult subjects (healthy or with respiratory disease - COPD) between 18 and 80 years of age, who will be enrolled in the pulmonary function laboratories of the participating hospitals, from among those listed above, who are attended to a functional respiratory examination.
  Interventions: Diagnostic Test: Mobile Web App

INTERVENTIONS:
Diagnostic Test: Mobile Web App — all participants will undergo an assessment of respiratory health by analyzing the sound of exhaled air recorded by the participant's mobile phone

SUMMARY:
Respiratory diseases are a common cause of mortality and disability at the worldwide and national levels. Many of them are characterized by underdiagnosis and diagnosis in advanced stages of the disease, and in most of them, forced spirometry is one of the fundamental tools to assess the diagnosis and seriousness of the disease.

To help in improving the detection of respiratory diseases and the understanding of the respiratory health of the general population, one possible solution would be to develop a mobile application that could assess respiratory health by using the sound signal of exhaled air recorded by a mobile microphone.

This project will aim to validate a mobile application (WebApp) for the detection of pulmonary function disorders. It is planned to recruit 267 subjects, with and without respiratory disease, who are attended in pulmonary function laboratories of 10 Spanish hospitals, to compare the sensitivity of this application in the diagnosis of pulmonary function disorders (either obstructive patterns or PRISm) versus the gold standard (spirometry). Ease of use and user satisfaction with the application will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with age range between 18 and 80 years old
* Signing the informed consent form
* Subjects scheduled for respiratory function tests at the pulmonary function laboratory for clinical reasons
* Having a cell phone and be willing to install the application

Exclusion Criteria:

* Contraindication to perform any of the protocol procedures
* Inability to answer the study questionnaires.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult subjects (healthy or with respiratory disease - COPD) between 18 and 80 years of age, who will be enrolled in the pulmonary function laboratories of the participating hospitals, from among those listed above, who are attended to a functional respiratory examination.
Sampling Method: Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Main Outcome | At the time of assessment
  Proportion of lung function abnormalities (defined as FEV1/FVC<0.7 or LLN) detected with the mobile app

SECONDARY OUTCOMES:
Secondary Outcome | At the time of assessment
  To analize the diagnostic performance from web app to detect different lung function abnormalities
Secondary Outcome | At the time of assessment
  To evaluate concordancy between lung function estimates obtained with a mobile app and spirometers
Secondary Outcome | At the time of assessment
  Proportion of lung function abnormalities (defined as FVC <80% predicted or LLN) detected with the mobile app

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Undecided